CLINICAL TRIAL: NCT02046499
Title: A Randomized Trial Comparing Oxytocin and Oxytocin + Ergometrine for Prevention of Postpartum Haemorrhage at Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Leon Snyman, Principal Specialist, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PPH Prevention Trial
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Prevention of Post Partum Haemorrhage
Keywords: Prevention, post partum haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; syntometrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin arm (Active Comparator): Oxytocin alone administered which is current standard of care
  Interventions: Drug: Oxytocin
- Oxytocin + syntometrine (Experimental): Oxytocin plus syntometrine administered
  Interventions: Drug: Oxytocin ergometrine

INTERVENTIONS:
Drug: Oxytocin — Oxytocin will be administered intravenously as per standard protocol
  Arms: Oxytocin arm
Drug: Oxytocin ergometrine — Oxytocin ergometrine will be administered intra-musculalry
  Other Names: Syntometrine
  Arms: Oxytocin + syntometrine

SUMMARY:
This is a randomized trial comparing oxytocin versus oxytocin + syntometrine in the prevention of post partum haemorrhage in patients undergoing caesarean section

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women delivering by caesarean section older than 18 years willing and able to give informed consent

Exclusion Criteria:

* • Women not willing or women not able to provide consent

  * Women who have a classical caesarean section
  * Women younger than 18 years of age
  * Women with any of the following conditions will be excluded (ergometrine contra-indicated in patients with these conditions).
  * Pre- eclampsia
  * Eclampsia,
  * Uncontrolled hypertension (hypertension defined as systolic blood pressure more than 140 mm Hg and diastolic blood pressure more than 90 mm Hg)
  * Any cardiac lesion
  * Impaired liver function
  * Impaired kidney function
  * Hypersensitivity to any of the active ingredients of the preparations that will be used (Syntometrine® or Syntocinon®)
  * Occlusive vascular disease
  * Autoimmune vasculitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-09-30 (Actual)

PRIMARY OUTCOMES:
Blood loss | 60 minutes
  Estimated blood loss at caesarean section

SECONDARY OUTCOMES:
Side effects of oxytocin compared to oxytocin + ergometrine | 24 hours
  Compare side effects experienced by women administered oxytocin compared to oxytocin plus ergometrine
Need for additional uterotonics | 60 minutes
  To determine the need for additional uterotonics to treat post partum haemorrhage
Number of units blood transfused | 24 hours
  Compare the number of units blood required for transfusion between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Leon C Snyman, MbChB MMed, Principal Investigator — Department Obstetrics & Gynaecology, University of Pretoria, South Africa
Locations (1):
- Kalafong Academic Hospital, Pretoria, Gauteng, South Africa